CLINICAL TRIAL: NCT05059197
Title: Evaluation of Skin Health Improvement and Safety in AP Collagen Peptide: Randomized, Double-blind, Placebo-controlled
Brief Title: Efficacy and Safety of AP Collagen Peptide on the Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PNK-20D21-FF1R
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-09

CONDITIONS: Dry Skin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AP collagen peptide (Experimental): Each subject takes one active bottle per day for 12 weeks. Each bottle contains AP collagen 1000 mg
  Interventions: Dietary Supplement: AP collagen peptide
- Placebo (Placebo Comparator): Each subject takes one active bottle per day for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: AP collagen peptide — Health functional food
  Arms: AP collagen peptide
Dietary Supplement: Placebo — placebo
  Arms: Placebo

SUMMARY:
This double-blinded, randomized, placebo-controlled study aimed to evaluate the efficacy and safety of AP collagen peptides (APCP) containing 3% Glycine-Proline-Hydroxyproline (GPH) on improving skin health. Subjects with dried skin were randomly assigned to receive placebo or APCP once daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Those whose eye wrinkles are Grade 3 or higher in the visual evaluation
* Those whose moisture retention in both cheeks measured by Corneometer® is 49 A.U. or less
* A person who has agreed to participate in this human application test before the start of the human application test and filled out the Informed Consent Form

Exclusion Criteria:

* Those with skin diseases such as atopic dermatitis and psoriasis
* Those who are sensitive to or allergic to the food ingredients for this trial foods
* Those with skin abnormalities such as spots, acne, erythema, and hypersensitive skin at the test site
* People who take diet pills (absorbent and antidepressants, appetite suppressants, etc.) and contraceptives or hormones or diuretics within one month based on visit1
* Those who have used functional cosmetics for wrinkle improvement, highly moisturizing cosmetics, or skincare devices within 2 weeks of visit 1
* A person who used steroid-containing outer skin for more than one month to treat skin diseases
* A person who has received chemical and physical treatment (pattern, epidermis, lasers, procedures, etc.) in the test area within six months prior to the start of the test
* Visit 1 A person who has participated in other interventional clinical tests (including human application tests) within one month of the standard or plans to participate in other interventional clinical tests (including human application tests) after the start of this human application test
* A person who judges that the tester is inappropriate for this test

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in epidermal hydration | Baseline, 12 week
  skin hydration measured by MoistureMeter-D compact

SECONDARY OUTCOMES:
Change from baseline in skin roughness (texture) | Baseline, 12 week
  skin roughness measured by PRIMOS
Change from baseline in skin gloss | Baseline, 12 week
  skin roughness measured by Skinglossmeter
Change from baseline in stratum corneum condition | Baseline, 12 week
  stripped using 10 tape strips (D-Squame) and measured by VisioScan
Change of Ceramides in stratum corneum | Baseline, 12 week
  ultra-performance liquid chromatography system etc.
Change of Natural moisturizing factor in stratum corneum | Baseline, 12 week
  Ultra-performance liquid chromatography system etc.
Change from baseline in TEWL | Baseline, 12 week
  Transepidermal water loss measured by vapometer

CONTACTS AND LOCATIONS:
Overall Officials: Hae Kwang Lee, PhD, Principal Investigator — P&K Skin Research Center
Locations (1):
- P&K Skin Research Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No